CLINICAL TRIAL: NCT00640302
Title: A Prospective Study to Examine the Effectiveness and Safety of Neuraminidase Inhibitors in Index Cases With Presumed Pandemic Influenza Infection
Brief Title: A Prospective Study to Examine the Effectiveness and Safety of Neuraminidase Inhibitors in Index Cases With Presumed Pandemic Influenza
Acronym: PIPET A
Status: Withdrawn | Type: Observational
Sponsor: Kirby Institute (Other Government)
Collaborators: National Health and Medical Research Council, Australia (Other)
Responsible Party: Associate Professor Sean Emery, The National Centre in HIV Epidemiology and Clinical Research
Other Study IDs: PIPET A
Record Dates: First submitted 2008-03-16; First posted 2008-03-21 (Estimated); Last update posted 2012-04-24 (Estimated); Status verified 2012-04

CONDITIONS: Pandemic Influenza
Keywords: Index cases; pandemic influenza; influenza A; H5N1 virus

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Patients will be asked to provide a blood sample and an appropriate respiratory tract sample. As a minimum, we will collect a combined nose and throat sample.
  A further respiratory tract swab will be collected on day 5 (range 5-10) and stored for future use. Index case follow-up will include an assessment and respiratory tract specimen and blood sample 14 days after informed consent. A final assessment for outcomes (including a blood sample) will occur approximately one month after enrolment.
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- PIPET A: Patients presenting at study sites with the recognised clinical case definition for pandemic influenza (to be distributed by State and Commonwealth Departments of Health when first clinical case occurs) will be eligible to be enrolled on the study. Informed consent to participate in the study will be sought including parental/guardian consent for minors and presumed consent for adults who are incapacitated (consistent with NHMRC requirements).

SUMMARY:
This aim of this project is to evaluate the efficacy of neuraminidase inhibitors in patients who have a clinical diagnosis of pandemic influenza infection. The study is observational only. The primary measure used in this study will be mortality. Symptom severity and duration, treatment limiting side effects, demographic information and resistance will also be examined. This project will commence upon pandemic influenza being declared in Australia, Hong Kong or Singapore. Data will be analysed as quickly as possible to help inform the continued use of neuraminidase inhibitor therapy as a cornerstone of the public health agency response to pandemic influenza.

DETAILED DESCRIPTION:
The aim of this study is to describe treatment outcomes in patients infected with pandemic influenza (the most likely case being a version of the influenza A H5N1 virus) including overall survival, the incidence and duration of hospitalization, the resolution of protocol specified symptoms, the incidence and the severity of treatment limiting side effects in treated patients. This study will also describe the sequelae of influenza in infected patients including transmission to other persons, associations between baseline data and treatment outcomes and drug resistance. A repository of biological samples will also be created to examine virological and immunological concepts relating to pandemic influenza.

It is an open label prospective cohort study. Patients presenting at study sites with the recognised clinical case definition for pandemic influenza (to be distributed by State and Commonwealth Departments of Health when first clinical case occurs) will be eligible to be enrolled on the study. Informed consent to participate in the study will be sought including parental/guardian consent for minors and presumed consent for adults who are incapacitated (consistent with NHMRC requirements).

ELIGIBILITY:
Inclusion Criteria:

* Clinical diagnosis of pandemic influenza (consistent with the applicable clinical case definition)
* Provision of written informed consent or equivalent
* Intention to commence treatment with a neuraminidase inhibitor

Exclusion Criteria:

* none

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Patients presenting at study sites with the recognised clinical case definition for pandemic influenza (to be distributed by State and Commonwealth Departments of Health when first clinical case occurs).
Sampling Method: Non-Probability Sample
Enrollment: 0 (Actual)

PRIMARY OUTCOMES:
Mortality | One month

CONTACTS AND LOCATIONS:
Overall Officials: Dominic Dwyer, FRACP, FRCPA, MD, Principal Investigator — Westmead Hospital
Locations (8):
- Australia (8):
  - St Vincent's Hospital, Sydney, New South Wales
  - Prince of Wales Hospital, Sydney, New South Wales
  - Westmead Hospital, Sydney, New South Wales
  - Royal Brisbane Hospital, Brisbane, Queensland
  - Flinders Medical Centre, Adelaide, South Australia
  - Royal Adelaide Hospital, Adelaide, South Australia
  - The Alfred Hospital, Melbourne, Victoria
  - Royal Perth Hospital, Perth, Western Australia